CLINICAL TRIAL: NCT03436342
Title: Chemokine Receptor CXCR4-targeting Molecular Imaging for Metabolic Characterization of Multiple Myeloma and Lymphoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCHCXCR4
Record Dates: First submitted 2017-10-25; First posted 2018-02-19 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-06

CONDITIONS: Multiple Myeloma; Lymphoma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma | interventions — 68Ga-pentixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-Pentixafor, PET/CT (Experimental): Inject 68Ga-Pentixafor and then perform PET/CT scan.
  Interventions: Drug: 68Ga-Pentixafor

INTERVENTIONS:
Drug: 68Ga-Pentixafor — Intravenous injection of one dosage of 74-148 MBq (2-4 mCi) 68Ga-Pentixafor. Tracer doses of 68Ga-Pentixafor will be used to image lesions of MM and lymphoma by PET/CT.

SUMMARY:
Chemokine receptor CXCR4 was expressed in MM and lymphoma cells and CXCR4-targeting molecular imaging- 68Ga-Pentixafor PET/CT could be a promising technique to evaluate the extent of MM and lymphoma with higher accuracy. This prospective study is going to investigate whether metabolic characterization by 68Ga-Pentixafor PET/CT may be superior for diagnosis, risk stratification, and prognostic evaluation of MM and lymphoma.

DETAILED DESCRIPTION:
Multiple myeloma:

Multiple myeloma (MM) is characterized by the neoplastic proliferation of plasma cells producing a monoclonal immunoglobulin. The Durie and Salmon and ISS clinical staging system have been well-accepted as a practical way to evaluate MM tumor burden nowadays. But it is difficult to assess the accurate tumor involvement because of the significant heterogeneity characterizing this disease at multiple levels such as clinical presentation, biologic characteristics, treatment response, and clinical outcome. New imaging modalities such as 18F-FDG PET/CT has been used to improve the efficacy of this system in assessing the extent and severity of MM, but the diagnostic accuracy of 18F-FDG PET/CT decreased in lower proliferative MM cells and inflammation. Recent studies showed Chemokine receptor CXCR4 was expressed in MM cells and CXCR4-targeting molecular imaging- 68Ga-Pentixafor PET/CT could be a promising technique to evaluate the extent of MM with higher accuracy. This prospective study is going to investigate whether metabolic characterization by 68Ga-Pentixafor PET/CT may be superior for diagnosis, risk stratification, and prognostic evaluation of MM.

Lymphoma:

Lymphoma is a frequent cancer with high CXCR4 expression. According to the previous studies, 68Ga-pentixafor-PET seems to be a highly selective and specific method for the in vivo quantification of CXCR4 expression. Thus our study is going to investigate the value of 68Ga-pentixafor-PET/CT for the diagnosis，differentiation and pretherapeutic evaluation of CXCR4 expression in lymphoma.

ELIGIBILITY:
Inclusion criteria：

* suspected or confirmed untreated MM or lymphoma patients
* 18F-FDG PET/CT within two weeks
* signed written consent.

Exclusion criteria:

* pregnancy
* breastfeeding
* known allergy against Pentixafor
* any medical condition that in the opinion of the investigator,may significantly interfere with study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
SUVmax | through study completion, an average of 2 years
  SUVmax of focal lesions are measured on 68Ga-Pentixafor PET/CT. The SUVmax of the L3 vertebra is defined as the general marrow activity on the condition that there is no focally hypermetabolic disease.

SECONDARY OUTCOMES:
Diagnostic value | through study completion, an average of 2 years
  Diagnostic value of 68Ga-Pentixafor PET/CT for MM and lymphoma in comparison with 18F-FDG PET/CT.
Incidence of emergency events during the study | through study completion, an average of 2 years
  Incidence of emergency events during the study
Tumor burden assessement | through study completion, an average of 2 years
  Correlation between tumor burden assessed on 68Ga-Pentixafor PET/CT and the DS and ISS clinical staging system for MM.
Diagnostic value in special type of multiple myeloma | through study completion, an average of 2 years
  Diagnostic value of 68Ga-Pentixafor PET/CT in monoclonal gammopathy of unknown significance (MGUS) and smoldering multiple myeloma (SMM) from symptomatic MM.
CXCR4 expression and SUV | through study completion, an average of 2 years
  Correlation between CXCR4 expression and SUV in PET
Overall Survival | 1 year and 5 years after been diagnosed
  analysis of OS for patients receiving 68Ga-Pentixafor PET/CT
Disease Free Survival | 1 year and 5 years after been diagnosed
  analysis of DFS for patients receiving 68Ga-Pentixafor PET/CT
Disease Specific Survival | 1 year and 5 years after been diagnosed
  analysis of DSS for patients receiving 68Ga-Pentixafor PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Fang Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Department of Nuclear Medicine, Peking Union Medical College Hopital, Chinese Academy of Medical Science, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pan Q, Chen Z, Liu S, Zhang H, Feng J, Miao W, Li F, Cao X, Luo Y. Reduced splenic uptake of [68Ga]Ga-Pentixafor following first-line chemotherapy is associated with poor prognosis in patients with newly diagnosed multiple myeloma. EJNMMI Res. 2025 Jun 20;15(1):74. doi: 10.1186/s13550-025-01262-2. PMID 40540129
- [Derived] Pan Q, Cao X, Luo Y, Li J, Feng J, Li F. Chemokine receptor-4 targeted PET/CT with 68Ga-Pentixafor in assessment of newly diagnosed multiple myeloma: comparison to 18F-FDG PET/CT. Eur J Nucl Med Mol Imaging. 2020 Mar;47(3):537-546. doi: 10.1007/s00259-019-04605-z. Epub 2019 Nov 27. PMID 31776631